CLINICAL TRIAL: NCT01120431
Title: The INcreased Flow Utilizing Subcutaneously-Enabled Time-Motion (INFUSE-TM) Study: A Randomized, Open-label, Parallel-group, Multicenter Study Evaluating Efficacy and Time and Resources in the Emergency Department for Hylenex-facilitated Subcutaneous Rehydration Versus Oral Rehydration Therapy in Pediatric Patients With Mild to Moderate Dehydration
Brief Title: Efficacy and Time and Resources for Hylenex-facilitated SC Rehydration Versus ORT for Dehydrated Children in the Emergency Department (ED)
Acronym: INFUSE-TM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Strategic business decision (not related to safety or efficacy concerns)
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1838-008
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Dehydration
Keywords: dehydration; fluid therapy; hyaluronoglucosaminidase; hyaluronidase; hypodermoclysis; clysis; subcutaneous hydration; subcutaneous rehydration; hyaluronan; rHuPH20; pediatric; ORT
MeSH Terms: conditions — Dehydration | interventions — Fluid Therapy; Ringer's Lactate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral rehydration therapy (Active Comparator)
  Interventions: Other: Oral rehydration fluid
- hylenex-facilitated SC hydration (Experimental)
  Interventions: Drug: Isotonic hydration fluid and recombinant human hyaluronidase

INTERVENTIONS:
Other: Oral rehydration fluid — Oral electrolyte solution or other clinically acceptable oral rehydration fluid, 5 to 10 mL of offered with encouragement every 5 to 10 minutes
  Other Names: oral rehydration salts
  Arms: Oral rehydration therapy
Drug: Isotonic hydration fluid and recombinant human hyaluronidase — Single subcutaneous dose of 150 U recombinant human hyaluronidase, followed by infusion pump-delivered subcutaneous isotonic hydration fluid
  Other Names: hyelenx; rHuPH20; Lactated Ringer's solution; normal saline solution; 0.9% sodium chloride solution
  Arms: hylenex-facilitated SC hydration

SUMMARY:
The purpose is to evaluate the safety and efficacy as well as the time and resources needed in the ED setting to achieve rehydration in young pediatric subjects with mild to moderate dehydration using hylenex-facilitated SC rehydration versus oral rehydration therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and aged 2 months to 2 years
* Presenting to ED with mild or moderate dehydration
* Candidate for both parenteral and oral rehydration therapies
* Healthy, except for underlying etiology for dehydration
* Naive to ORT or having received attempted ORT at home for current occurrence of dehydration.
* Pre-dehydration body weight greater than 5th percentile for age

Exclusion Criteria:

* Severe dehydration
* Shock or a life-threatening situation
* Any condition precluding SC infusion or infusion site evaluation in all possible anatomical locations (upper back, anterior thighs, abdomen, other potential areas) for SC infusion
* Medical reason or condition precluding administration of ORT
* Indwelling IV catheter (except one intended only for laboratory sample collection) or anticipated need for IV therapy during the study
* Anticipated need for hospitalization(other than for rehydration)
* Known hypersensitivity to hyaluronidase or any other ingredient in the formulation of hylenex recombinant
* Known hyponatremia, hypernatremia or hypokalemia
* Medical condition likely to interfere with ability to fully complete protocol-specified interventions and assessments, or likely to prolong need for medical attention beyond that required for rehydration
* Participation in an investigational drug or device study within 30 days before participation in this study

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-05 (Estimated); Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Total resource utilization in the ED | 2 to 8 hours

SECONDARY OUTCOMES:
Rate of successful rehydration in the ED | 2 to 8 hours
  Clinical judgement of adequate hydration, and either: 1) stable or increased body weight or 2) urine production
Time to ED discharge | 2 to 8 hours
Amount of rehydration fluid administered | 2 to 8 hours
Global satisfaction and ease-of-use assessments by healthcare provider(s) and parent/caregiver | 2 to 8 hours
Occurrence of infusion site pain or other local reactions | 2 to 8 hours
Occurrence of other adverse events | 7 days
Vital signs | 2 to 8 hours
  Blood pressure, heart rate, respiratory rate, temperature

CONTACTS AND LOCATIONS:
Overall Officials: George Harb, MD, MPH, Study Director — Baxter Healthcare Corporation